CLINICAL TRIAL: NCT05332249
Title: Registry for Degenerative Spinal Disease
Brief Title: Registry for Degenerative Spinal Disease (RDSD)
Acronym: RDSD
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Degenerative registry
Record Dates: First submitted 2022-03-01; First posted 2022-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Degeneration Spine; Surgery
Keywords: Spine; Outcomes; Degeneration spine; Surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar: Patients undergo lumbar spinal surgery for degenerative lumbar spinal disease.
  Interventions: Procedure: Surgery
- Cervical: Patients undergo cervical spinal surgery for degenerative cervical spinal disease.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Patients who undergo spinal surgery for degenerative spinal disease

SUMMARY:
The outcome after spinal surgery is important and the evidence is critical to develop treatment. The purpose of this study is to make a prospective registry of database for further research.

DETAILED DESCRIPTION:
The outcome after spinal surgery is important and the evidence is critical to develop treatment. The purpose of this study is to make a prospective registry of database for further research.

Included patients Degenerative cervical spinal disease. Degenerative lumbar spinal disease.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative lumbar spinal disease.
* Degenerative Cervical spinal disease

Exclusion Criteria:

* combined progressive cancer disease

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are going to take surgery at Seoul National University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2050-12-30 (Estimated); Study Completion 2050-12-30 (Estimated)

PRIMARY OUTCOMES:
Disability index | 20 years
  Improve of disability index more than 30% from the baseline

SECONDARY OUTCOMES:
C7-sagittal vertical axis (C7-SVA) | 20 years
  Change of C7-SVA, quantative comparison between preoperation and postoperative year 20 years.
European quality of life questionnare _ 5 dimension (EQ-5D) | 20 years
  Improve of EQ-5D more than 30% from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chi Heon Kim, pf., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No